CLINICAL TRIAL: NCT00630812
Title: Long Term Administration of Inhaled Mannitol in Cystic Fibrosis- A Safety and Efficacy Study
Brief Title: Long Term Administration of Inhaled Mannitol in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syntara (Industry)
Collaborators: ethica Clinical Research Inc. (Industry); Europe: KasaConsult bvba, Hoegaarden, Belgium (Industry); Resolution Latin America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPM-CF-302
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mannitol; mucoactive
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): active treatment
  Interventions: Drug: inhaled mannitol
- B (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: inhaled mannitol — 400 mg BD for 26 + 26 weeks
  Arms: A
Drug: Placebo comparator — BD for 26 weeks followed by 26 weeks of inhaled mannitol in the open label phase
  Arms: B

SUMMARY:
The purpose of this study is to examine the efficacy and safety of 26 weeks treatment with inhaled mannitol in subjects with cystic fibrosis. Previous studies have demonstrated improvements in lung function, mucociliary clearance, changes in physical properties of mucus, 24 hour sputum weight and quality of life. The results of this study are to further investigate and confirm these findings in addition to examine the effect on antibiotic use and chest infections. It is hypothesised that inhaled mannitol will have beneficial effects compared to a control treatment. An open label phase of 26 weeks duration will follow the blinded 26 week phase. During the open label phase all subjects will receive active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent to participate in this study in accordance with local regulations
2. Have a confirmed diagnosis of cystic fibrosis (positive sweat chloride value ≥ 60 mEq/L) and/or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with the CF phenotype)
3. Be aged > 6 years old
4. Have FEV1 >40 % and < 90% predicted
5. Be able to perform all the techniques necessary to measure lung function

Exclusion Criteria:

1. Investigators, site personnel directly affiliated with this study, or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted.
2. Be considered "terminally ill" or eligible for lung transplantation
3. Have had a lung transplant
4. Be using nebulized hypertonic saline in the 4 weeks prior to visit 1
5. Have had a significant episode of hemoptysis (>60 mL) in the three months prior to enrolment
6. Have had a myocardial infarction in the three months prior to enrolment
7. Have had a cerebral vascular accident in the three months prior to enrolment
8. Have had major ocular surgery in the three months prior to enrolment
9. Have had major abdominal, chest or brain surgery in the three months prior to enrolment
10. Have a known cerebral, aortic or abdominal aneurysm
11. Be breast feeding or pregnant, or plan to become pregnant while in the study
12. Be using an unreliable form of contraception (female subjects at risk of pregnancy only)
13. Be participating in another investigative drug study, parallel to, or within 4 weeks of visit 0
14. Have a known allergy to mannitol
15. Be using beta blockers
16. Have uncontrolled hypertension - systolic BP > 190 and / or diastolic BP > 100
17. Have a condition or be in a situation which in the Investigator's opinion may put the subject at significant risk, may confound results or may interfere significantly with the patient's participation in the study
18. Be 'Mannitol Tolerance Test positive'

    -

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moira L Aitken, MD, Principal Investigator — University of Washington Medical Centre, Seattle WA
Locations (53):
- United States (28):
  - University of Arizona, Tucson, Arizona
  - Central Connecticut Cystic Fibrosis Center, Hartford, Connecticut
  - Nemours Childrens Clinic, Jacksonville, Florida
  - Batchelor Children's Research Institute - University of Miami, Miami, Florida
  - Nemours Children's Clinic Orlando, Orlando, Florida
  - St Lukes CF Center of Idaho, Idaho City, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Maine Pediatric Specialty Group, Portland, Maine
  - John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Nebraska Medical Center - Nebraska Regional CF Center, Omaha, Nebraska
  - Women and Childrens Hospital of Buffalo, Buffalo, New York
  - The Toledo Hospital and Toledo Childrens Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of SC, Charleston, South Carolina
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - Le Bonheur Children's Medical Center, Memphis, Tennessee
  - Children's Chest Associates of Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Christus Santa Rosa Children's Hospital Cystic Fibrosis Center, San Antonio, Texas
  - Pediatric Research, VCU Medical Centre, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington medical centre, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (8):
  - Hospital Interzonal Dr Jose Penna Bahia Blanca, Bahía Blanca, Buenos Aires
  - Hospital de Ninos Dr Ricardo Gutierrez, Pediatria, CABA, Buenos Aires
  - Hospital Gral. de Ninos Pedro de Elizalde, Ciudad Autonoma, Buenos Aires
  - Hospital de Ninos Superiora Sor Maria Ludovica de La Plata, La Plata, Buenos Aires
  - Hospital Pediatrico Dr Humberto J Notti, Villa Nueva, Mendoza Province
  - Atención Integral en Reumatologia (AIR), Buenos Aires
  - Clinica Universitaria Privada Reina Fabiola - Universidad Cotolica de Cordoba, Córdoba
  - Hospital de Ninos del la Santisima Trinidad, Córdoba
- Belgium (4):
  - Pediatrics Respiratory Medicine, Edegem, Antwerpen
  - Hopital Universitaire Reine Fabiola, Brussels, Brussels Capital
  - UZ Brussel Laarbeeklan 101, Brussels
  - UZ Gasthuisberg, Leuven
- Canada (3):
  - Foothills medical center, Calgary, Alberta
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - The Children's Asthma Clinic, London, Ontario
- France (6):
  - Hopital Mere-Enfant, Nantes, Cedex
  - Hopital Andre Mignot, Le Chesnay, Cedix
  - Hopital Jeanne de Flandre, Lille, Lille
  - Hopital Femme-Mere-Enfents, Bron, Lyon
  - Hopital de Hautepierre, Strasbourg, Strasbourg
  - Hopital Robert Debre, Paris
- Germany (3):
  - University of Munich Medizinischen Klinik Innenstadt, München
  - Universitats Kinderklinik Tubungen Wurzburg, Tübingen
  - Universitats Kinderklinik Wurzburg, Würzburg
- Academic Medical Centre, Amsterdam, Netherlands

REFERENCES:
- [Background] Daviskas E, Anderson SD. Hyperosmolar agents and clearance of mucus in the diseased airway. J Aerosol Med. 2006 Spring;19(1):100-9. doi: 10.1089/jam.2006.19.100. PMID 16551221
- [Background] Daviskas E, Anderson SD, Gomes K, Briffa P, Cochrane B, Chan HK, Young IH, Rubin BK. Inhaled mannitol for the treatment of mucociliary dysfunction in patients with bronchiectasis: effect on lung function, health status and sputum. Respirology. 2005 Jan;10(1):46-56. doi: 10.1111/j.1440-1843.2005.00659.x. PMID 15691238
- [Background] Daviskas E, Robinson M, Anderson SD, Bye PT. Osmotic stimuli increase clearance of mucus in patients with mucociliary dysfunction. J Aerosol Med. 2002 Fall;15(3):331-41. doi: 10.1089/089426802760292681. PMID 12396422
- [Background] Robinson M, Bye PT. Mucociliary clearance in cystic fibrosis. Pediatr Pulmonol. 2002 Apr;33(4):293-306. doi: 10.1002/ppul.10079. PMID 11921459
- [Background] Daviskas E, Anderson SD, Eberl S, Chan HK, Young IH. The 24-h effect of mannitol on the clearance of mucus in patients with bronchiectasis. Chest. 2001 Feb;119(2):414-21. doi: 10.1378/chest.119.2.414. PMID 11171717
- [Background] Robinson M, Daviskas E, Eberl S, Baker J, Chan HK, Anderson SD, Bye PT. The effect of inhaled mannitol on bronchial mucus clearance in cystic fibrosis patients: a pilot study. Eur Respir J. 1999 Sep;14(3):678-85. doi: 10.1034/j.1399-3003.1999.14c30.x. PMID 10543292
- [Background] Daviskas E, Anderson SD, Eberl S, Chan HK, Bautovich G. Inhalation of dry powder mannitol improves clearance of mucus in patients with bronchiectasis. Am J Respir Crit Care Med. 1999 Jun;159(6):1843-8. doi: 10.1164/ajrccm.159.6.9809074. PMID 10351929
- [Background] Daviskas E, Anderson SD, Brannan JD, Chan HK, Eberl S, Bautovich G. Inhalation of dry-powder mannitol increases mucociliary clearance. Eur Respir J. 1997 Nov;10(11):2449-54. doi: 10.1183/09031936.97.10112449. PMID 9426077
- [Background] Jaques A, Daviskas E, Turton JA, McKay K, Cooper P, Stirling RG, Robertson CF, Bye PTP, LeSouef PN, Shadbolt B, Anderson SD, Charlton B. Inhaled mannitol improves lung function in cystic fibrosis. Chest. 2008 Jun;133(6):1388-1396. doi: 10.1378/chest.07-2294. Epub 2008 Mar 13. PMID 18339790
- [Derived] Nevitt SJ, Thornton J, Murray CS, Dwyer T. Inhaled mannitol for cystic fibrosis. Cochrane Database Syst Rev. 2020 May 1;5(5):CD008649. doi: 10.1002/14651858.CD008649.pub4. PMID 32358807
- [Derived] Aitken ML, Bellon G, De Boeck K, Flume PA, Fox HG, Geller DE, Haarman EG, Hebestreit HU, Lapey A, Schou IM, Zuckerman JB, Charlton B; CF302 Investigators. Long-term inhaled dry powder mannitol in cystic fibrosis: an international randomized study. Am J Respir Crit Care Med. 2012 Mar 15;185(6):645-52. doi: 10.1164/rccm.201109-1666OC. Epub 2011 Dec 28. PMID 22198974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients underwent a mannitol tolerance test (MTT) to gauge tolerance to a test dose of mannitol. 318 patients were then randomised - only 305 of the randomised patients went on to receive a dose of study medication. Patients who did not start medication (13) were not included in the modified ITT population (mITT)
Groups:
- Mannitol 400mg: active treatment
  inhaled mannitol: 400 mg twice a day (BD) for 26 + 26 weeks
- Control: Control (40mg inhaled mannitol) : BD for 26 weeks followed by 26 weeks of inhaled mannitol in the open label phase
Period: Randomisation to First Dose
Arm/Group | Mannitol 400mg | Control
Started | 192 | 126
Completed | 184 | 121
Not Completed | 8 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 4 | 1
Period: Double Blind Treatment Period
Arm/Group | Mannitol 400mg | Control
Started (Randomised and received first dose (mITT population). Patients not starting treatment are excluded) | 184 | 121
Completed | 153 | 107
Not Completed | 31 | 14
Not completed — Adverse Event | 13 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Wanted to take drug in non-protocol way | 1 | 0
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomised and Treated (mITT)
Groups:
- Mannitol 400mg: active treatment
  inhaled mannitol: 400 mg BD for 26 + 26 weeks
- Total: Total of all reporting groups
Arm/Group | Mannitol 400mg | Control | Total
Number analyzed (Participants) | 184 | 121 | 305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91 | 63 | 154
  Between 18 and 65 years | 93 | 58 | 151
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 58 | 148
  Male | 94 | 63 | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 182 | 119 | 301
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 9 | 20
  Argentina | 48 | 32 | 80
  Netherlands | 2 | 2 | 4
  Belgium | 10 | 6 | 16
  United States | 85 | 54 | 139
  France | 14 | 9 | 23
  Germany | 14 | 9 | 23
Hospitalisations in year prior to study participation [Count of Participants; unit: Participants]
  0 hospitalisations | 114 | 76 | 190
  1 hospitalisation | 41 | 30 | 71
  2 hospitalisations | 21 | 9 | 30
  3 hospitalisations | 4 | 4 | 8
  >3 hospitalisations | 4 | 2 | 6
Pulmonary exacerbations in year prior to study participation [Count of Participants; unit: Participants]
  0 exacerbations | 104 | 74 | 178
  1 exacerbation | 45 | 28 | 73
  2 exacerbations | 26 | 14 | 40
  3 exacerbations | 4 | 3 | 7
  >3 exacerbations | 5 | 2 | 7
CF mutation [Count of Participants; unit: Participants] — Cystic Fibrosis (CF) mutation
  Participants
    Both deltaF508 | 77 | 45 | 122
    One deltaF508 | 57 | 52 | 109
    At least one other known mutation | 15 | 5 | 20
    Both unknown | 35 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute FEV1 From Baseline Over 26 Weeks
Description: Change from baseline in forced expiratory volume at one second (FEV1) averaged over 26 weeks (measured at 6,14 and 26 weeks) The mean absolute change from baseline FEV1 (mL) over 26 weeks (measured at week 6, 14 and 26) will be compared between the two treatment groups with a REML (restricted maximum likelihood) based repeated measures approach.Least square means presented are for the average change over the 6, 14, and 26 week visits.
Time Frame: 26 weeks
Population: mITT (modified intent to treat) - patients randomised and treated with at least one dose of study medication)
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
mL | 106.53 [62.43 to 150.62] | 52.38 [2.09 to 102.68]
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Net) = 54.14, 95% CI 2-sided [-1.97 to 110.26]
Statistical Analysis 2: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.041, Regression, Logistic — Response defined as change of >=100mL at week 26; 45.7% response on Mannitol 400mg, 35.5% on Control; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.02 to 2.80]

2. Secondary Outcome: Change in FEV1 From Baseline Over 26 Weeks - Dornase Users
Description: In the subset of dornase users, the mean absolute change from baseline FEV1 (mL) averaged over 26 weeks (measured at week 6, 14 and 26) will be compared between the two treatment groups with a REML (restricted maximum likelihood) based repeated measures approach. Least square means presented are for the average change over the 6, 14, and 26 week visits.
  Change from baseline over 26 weeks (measured at 6,14, 26 weeks) in subset of dornase users
Time Frame: 26 weeks
Population: Note these are subset of dornase users - effect in dornase users was estimated using a model fitted using data from all patients
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 137 | 92
mL | 78.60 [27.64 to 129.56] | 35.11 [-20.99 to 91.21]
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.177, Mixed Models Analysis; Mean Difference (Net) = 43.49, 95% CI 2-sided [-19.8 to 106.78]

3. Secondary Outcome: Rate of Protocol Defined Pulmonary Exacerbations (PDPE)
Description: Exacerbations treated with IV antibiotics and with at least 4 signs and symptoms according to Fuchs criteria (1994). Summary table presents the number with 0, 1,2 and 3 PDPEs during the 26 week treatment period.
Time Frame: 26 weeks
Population: mITT (randomised and treated)
Measure: Count of Participants; unit: Participants
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
Participants
  With 1 PDPE | 21 | 18
  With 2 PDPE | 6 | 4
  With 3 PDPE | 1 | 1
  No PDPEs | 156 | 98
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.520, Poisson regression; Offset of the natural logarithm of follow-up time; Rate ratio = 0.85, 95% CI 2-sided [0.51 to 1.41]

4. Secondary Outcome: Hospitalisations Associated With Protocol Defined Pulmonary Exacerbations (PDPEs)
Description: The number of hospitalisations is summarised and then the rate per person is analysed.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
Participants
  0 hospitalisations | 162 | 102
  1 hospitalisation | 18 | 14
  2 hospitalisations | 3 | 5
  3 hospitalisations | 1 | 0
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.328, Poisson regression; Offset of the natural logarithm of follow-up time; Rate ratio = 0.75, 95% CI 2-sided [0.42 to 1.33]

5. Secondary Outcome: Antibiotic Use Associated With PDPEs
Description: Number of courses per person in the 26 week period is summarised and then the rate per person analysed.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
Participants
  0 courses | 156 | 98
  1 course | 22 | 19
  2 courses | 5 | 2
  3 courses | 1 | 2
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.368, Poisson regression; Rate ratio = 0.89, 95% CI 2-sided [0.69 to 1.15]

6. Secondary Outcome: Absolute Change in FEV1 Percent Predicted at 26 Weeks
Description: Change from baseline at 26 weeks in FEV1 percent predicted with BOCF for those with missing values at week 26
Time Frame: 26 weeks
Population: Baseline Observation carried forward (BOCF) implemented for those with missing values at visit 4
Measure: Least Squares Mean (95% Confidence Interval); unit: % of predicted
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
% of predicted | 3.14 [1.49 to 4.78] | 0.72 [-1.18 to 2.62]
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.024, ANCOVA; Mean Difference (Net) = 2.42, 95% CI 2-sided [0.33 to 4.51]

7. Secondary Outcome: Change in FVC (mL) Across 26 Weeks
Description: Change from baseline in forced vital capacity (FVC) across 26 weeks (measured at 6,14 and 26 weeks)
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
mL | 136.33 [88.54 to 184.11] | 64.98 [10.58 to 119.37]
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Net) = 71.35, 95% CI 2-sided [10.57 to 132.13]

8. Secondary Outcome: Change From Baseline FEF25-75 (mL/s) Over 26 Weeks
Description: Change from baseline in forced expiratory flow at 25-75% of forced vital capacity (FEF25-75) (mL/s) averaged over 26 weeks (measured at 6,14 and 26 weeks) The mean absolute change from baseline over 26 weeks (measured at week 6, 14 and 26) was compared between the two treatment groups with a REML (restricted maximum likelihood) based repeated measures approach. Least square means presented are for the average change over the 6, 14, and 26 week visits.
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/s
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 184 | 121
mL/s | 84.65 [6.66 to 162.63] | 50.31 [-38.24 to 138.86]
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Net) = 34.34, 95% CI 2-sided [-63.47 to 132.14]

9. Secondary Outcome: Sputum Weight at Baseline in Response to First Dose of Treatment
Description: Sputum was collected during and for 30 minutes following the administration of the first dose of study treatment.
Time Frame: up to 30 mins after first dose of trial treatment
Population: Patients randomised and treated who have sputum weight results available.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Mannitol 400mg | Control
Number analyzed (Participants) | 180 | 114
g | 4.9 (6.18) | 3.5 (4.40)
Statistical Analysis 1: Comparison: Mannitol 400mg vs Control; Test type: Superiority; p = 0.042, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Safety information reported is for the 26 week double blind period only
Arm/Group | Mannitol 400mg | Control
All-Cause Mortality (participants affected / at risk) | 0/184 | 1/121
Serious Adverse Events (participants affected / at risk) | 31/184 | 30/121
Other Adverse Events (participants affected / at risk) | 165/184 | 106/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mannitol 400mg (N=184) | Control (N=121)
Condition Aggravated (General disorders) | 27 | 20 — pulmonary exacerbations were coded to condition aggravated
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Acute tonsillitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mannitol 400mg (N=184) | Control (N=121)
Condition Aggravated (General disorders) | 57 | 41 — Pulmonary Exacerbations were coded to condition aggravated
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 16
Headache (Nervous system disorders) | 26 | 22
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Pyrexia (General disorders) | 17 | 13
Abdominal pain (Gastrointestinal disorders) | 14 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Nasopharyngitis (Infections and infestations) | 11 | 6
Upper respiratory tract infection (Infections and infestations) | 10 | 11
Sinusitis (Infections and infestations) | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No